CLINICAL TRIAL: NCT02347007
Title: Impact of Almond Supplementation, Relative to a Low-fat, High Carbohydrate Control, on Body Composition in Overweight and Obese Black and Hispanic Adults
Brief Title: Impact of Almond Supplementation on Body Composition in Overweight/Obese Minority Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAN4353
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Overweight; Fatty Liver; Metabolic Syndrome X
Keywords: Obesity; Overweight; Body Weight; Cardiovascular Diseases; Cholesterol; Almonds; Visceral Adiposity; Quality of Life; Hispanic Americans; African Continental Ancestry Group; Metabolic Syndrome X
MeSH Terms: conditions — Obesity; Overweight; Fatty Liver; Metabolic Syndrome; Body Weight; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Almond (Experimental)
  Interventions: Dietary Supplement: Almond
- Cereal Bar (Active Comparator)
  Interventions: Dietary Supplement: Cereal Bar

INTERVENTIONS:
Dietary Supplement: Almond — Participants will be randomized to consume approximately 17.5% of their estimated energy requirements from almonds daily for 24 weeks. Prescribed energy requirements will be determined for each participant individually using the Mifflin St Jeor Equation equation with an activity factor of 1.3. Participants will be asked to consume half of their daily almond supplement as a mid-afternoon snack and the rest at a meal of their choice.
  Arms: Almond
Dietary Supplement: Cereal Bar — Participants will be randomized to consume approximately 17.5% of their estimated energy requirements from cereal bars daily for 24 weeks. Prescribed energy requirements will be determined for each participant individually using the Mifflin St Jeor Equation equation with an activity factor of 1.3. Participants will be asked to consume half of their daily cereal bar supplement as a mid-afternoon snack and the rest at a meal of their choice.
  Arms: Cereal Bar

SUMMARY:
The purpose of this study is to determine whether introducing almonds into the diet of overweight and obese Blacks and Hispanics improves body composition, decreases liver fat, and lowers cardiovascular disease profile.

DETAILED DESCRIPTION:
The study is a randomized, controlled study aimed at testing whether almonds, consumed within a free-living, self-selected diet, improve body composition and liver fat, relative to a low-fat/high-carbohydrate cereal bar (LF-HC) in overweight and obese Blacks and Hispanics. A secondary aim is to determine whether almond consumption will lead to an overall lower CVD risk profile.

Participants will be randomized to consume approximately 17.5% of their estimated energy requirements from almonds daily (2-3 oz) or a high-carbohydrate cereal bar (2 g of fat or less per 100 kcal) providing an equivalent amount of calories. Prescribed energy requirements will be determined for each participant individually using the Mifflin St Jeor Equation equation with an activity factor of 1.3. Participants will be asked to consume half of their food supplement as a mid-afternoon snack and the rest at a meal of their choice.

At the baseline visit, participants will be given a 2-week supply of their allocated food supplement and will obtain additional supplies at bi-weekly visits for the first 8 weeks. After the week 8 visit, participants will be given monthly rations of their food supplement, either almonds or LF-HC cereal bar, and will be asked to come to research center every 4 weeks to obtain their next supply. At those visits, body weight and blood pressure will be measured and participants will turn in weekly dietary diaries, reporting their supplement intake. Participants will also receive one random phone call every 4 weeks to provide a 24-h recall. This recall will be used as an index of dietary quality but also as a compliance check with dietary supplements. In addition, 3-day food records will be collected prior to the start of the study and during the final week to assess any dietary changes due to the intervention. A food frequency questionnaire will also be administered at screening and endpoint of the study. This food-frequency questionnaire will target nut consumption.

At the end of the study, intention to continue eating almonds or a low-fat diet will be assessed using questions adapted from de Bruijn et al. Participants in the almond group will be asked the following questions: (1) "I intend to include almonds in my diet" (+2 = yes, definitely; -2 = no, definitely); (2) "How certain are you that you will include almonds in your diet?" (+2 = very certain; -2 = very uncertain); (3) "Including almonds in my diet is" (instrumental attitude: +3 = healthy; -3 = unhealthy; affective attitude: +3 = pleasant; -3 = unpleasant); (4) "I find including almonds in my diet" (perceived behavioral control: +3 = easy; -3 = difficult). Corresponding questions for the control group will replace "include almonds" with "reduce the amount of fat". Participants will be called 4 weeks later to obtain information on their actual almond and fat intakes by questionnaire and 24-h recall.

ELIGIBILITY:
Inclusion Criteria:

* Black and/or Hispanic
* Body Mass Index (BMI) 25-35 kg/m^2
* Weight stable (+/- 2.5 kg) for at least 3 months prior to screening
* Body weight less than 300 pounds
* Adherence to an acceptable form of contraception (for women)
* If taking medicine, dose must have been stable before study; must remain on same medication and dose throughout study.

Exclusion Criteria:

* Diabetes
* Uncontrolled hypertension (high blood pressure)
* Cardiovascular disease
* Weight loss attempted in past 3 months
* Eating disorder
* Stroke, seizure disorder, or significant neurological disease
* Unstable of uncontrolled medical illness including active malignancies within past 5 years
* Untreated or unstable hypothyroidism
* Hyperthyroidism
* Diagnosis of psychoses, bipolar disorder, major depression, severe personality disorder; history of suicidal tendencies
* Alcohol or substance abuse in the past 6 months
* Pregnant, planning pregnancy in the next 6 months, or breast-feeding
* Participating or planning to participate in a commercial diet or behavior modification program (ex: Weight Watchers)
* Allergy or sensitivity to wheat/grain products or nuts
* Gastrointestinal disorder.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in body Composition | Baseline and endpoint visits (Weeks 0 and 24)
  MRI will be used to provide information on total adipose tissue and all adipose tissue sub-compartments: visceral, subcutaneous, intermuscular.
Change in liver Fat | Baseline and endpoint visits (weeks 0 and 24)
  MRS will be used to provide information on liver adiposity.

SECONDARY OUTCOMES:
Change in cardio-metabolic risk profile | Baseline, midpoint, and endpoint visits (weeks 0, 12, and 24)
  Blood draw and analyses will be used to measure total and low-density lipoprotein cholesterol, triglycerides, high-density lipoprotein cholesterol, glucose, insulin, and inflammatory markers.
Change in brain-derived neutrophic factor (BDNF) | Baseline, midpoint, and endpoint visits (weeks 0, 12, and 24)
  Blood draw and analyses will be used measure BDNF.
Change in quality of life | Baseline and endpoint visits (weeks 0 and 24)
  SF-36 questionnaire will be used to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D., Principal Investigator — College of Physicians & Surgeons, Columbia University
Locations (1):
- New York Nutrition Obesity Research Center, New York, New York, United States